CLINICAL TRIAL: NCT05837143
Title: An Exploratory Clinical Study of JV001 in the Treatment of Patients With Heart Failure Due to Dilated Cardiomyopathy (Telomere Recapping to Restore Mitochondrial Biogenesis Study for Dilated Cardiomyopathy)
Brief Title: Myocardial Telomere Recapping Study for Dilated Cardiomyopathy
Acronym: MERCURY-DCM
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai Juvensis Therapeutics Biotechnology Company Limited (Unknown)
Responsible Party: Principal Investigator, Wei Han, Director, Head of Heart Failure Unit, Principal Investigator, Clinical Professor, Shanghai East Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JV001-02
Record Dates: First submitted 2023-03-24; First posted 2023-05-01 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Dilated Cardiomyopathy
Keywords: Adeno-associated virus; modTERT; Dilated Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Comparator: JV001 (Experimental): Subjects will receive a single intracoronary infusion of JV001 at a dose of 2×10^11vg/kg, and 6×10^11vg/kg.
  Interventions: Biological: JV001

INTERVENTIONS:
Biological: JV001 — JV001 (AAV9/modTERT) will be delivered by a percutaneous method in the catheter laboratory. Dose: 2×10^11vg/kg，or 6×10^11vg/kg.

SUMMARY:
The aim of this study is to determine the safety and feasibility of giving an adeno-associated viral vector expressing a modified telomerase protein (TERT), driven by cardiac troponin T promoter (AAV9-cTnT-modTERT), to 12 dilated cardiomyopathic patients.

DETAILED DESCRIPTION:
It is an open-label, 6+6 design study involving two dosages ( 2×10^11vg/kg, and 6×10^11vg/kg) aimed to explore the safety, pharmacokinetics, immunology, and preliminary efficacy of JV001.

ELIGIBILITY:
Inclusion Criteria:

* DCM≥1year;
* NYHA II-IV;
* LVEF ≤35%；
* Received maximally tolerated guideline-directed medical therapy (GDMT) for at least 3 months before enrollment with persistent heart failure; or unable to tolerate standardized pharmacotherapy recommended by guidelines (according to clinical data), but in which investigators assessed participants who could benefit from the study drug; or hospitalized for heart failure more than 2 times within 1 year and requiring intravenous diuretic therapy, while the condition is stable for more than 2 weeks;
* Have the ability to understand and voluntarily sign informed consent before the trial, and be able to complete the study in accordance with the requirements of the trial protocol;
* Male or female: (1) male subjects must agree to use contraception for at least 6 months after treatment visit; (2) the female subjects were not pregnant or breastfeeding; (3) Females of childbearing potential agree to comply with contraceptive guidance for at least 6 months after administration (see Appendix 1)

Exclusion Criteria:

* Patients with heart failure caused by heart diseases other than dilated cardiomyopathy (including but not limited to severe valvular heart disease, hyperthyroidism, congenital heart disease, acute viral myocarditis, acute coronary syndrome, hypertrophic obstructive cardiomyopathy, pericardial disease, myocardial amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or left ventricular aneurysm).
* Coronary angiography has a degree of narrowing of the left main coronary artery (LM), left anterior descending branch (LAD), left circumflex branch (LCX) or right coronary artery (RCA) > 50%.
* Uncontrolled arrhythmias that the investigator believes would affect this trial.
* Acute myocardial infarction within 6 months before screening
* Previous presence of subjects with immunological abnormalities that the investigators believe could affect this trial (including but not limited to congenital immunodeficiency, lupus erythematosus, primary vasculitis, systemic sclerosis, antiphospholipid syndrome, autoimmune liver disease, autoimmune thyroiditis).
* Those who have a history of tumor for less than 5 years or currently have a tumor, or those who have precancerous lesions confirmed by pathological examination (including but not limited to breast ductal carcinoma in situ, cervical dysplasia, etc.)
* Known progress liver disease (active hepatitis A, chronic hepatitis B or C virus infection, non-cardiogenic cirrhosis, etc.)
* Acute infection developed within 2 weeks prior to screening requiring intravenous antibiotic therapy, or current infection requiring anti-infective therapy.
* Those who have a history of disseminated herpes simplex infection or recurrent (> 1 times) or disseminated herpes zoster.
* Percutaneous coronary intervention (PCI), coronary bypass grafting (CABG), Implantable Cardioverter Defibrillator (ICD)/permanent pacemaker/Cardiac resynchronisation therapy (CRT) implantation, radiofrequency ablation, ventricular volume reduction, valve repair or plasty, intra-aortic balloon counterpulsation, passive restraint devices (e.g., CorCap™ cardiac support devices), cardiac assist device implantation, heart transplantation, or other cardiac surgery may be received within 3 months prior to screening or within 3 months after administration.
* Those who donated ≥ 400 mL of blood within 4 weeks prior to screening, or who had significant blood loss equivalent to at least 400 mL, or who received blood transfusions within 8 weeks.
* Subjects with contraindications for coronary angiography
* Contraindications for Magnetic Resonance Imaging (MRI) detection, including but not limited to: pacemaker, defibrillator, artificial heart valve, metal clip after aneurysm surgery, drug perfusion device implanted in the body, any electronic device implanted in the body (neurostimulator, bone growth stimulator), intravascular embolization steel ring, filter, ECG recording monitor, shrapnel or iron sand in the body, fixed steel plate and nails after fracture surgery, cochlear implant, intraocular metal foreign body, etc.; Claustrophobia, etc.
* Those who have a history of substance abuse within the past five years or have used drugs in the 3 months prior to the test.
* Are participating in other clinical trials, or have been completed less than 3 months after the end of other clinical trials.
* Abnormal liver function: ALT or AST > 3 times the upper limit of normal value (ULN).
* Abnormal renal function: glomerular filtration rate < 30 mL/min or dialysis-dependent.
* Hematologic disorders: thrombocytopenia is defined as <50,000 platelets/μL within 30 days prior to screening; Anaemia is defined as haemoglobin <10 g/dL within 30 days prior to screening or dependence on blood transfusion; Neutropenia is defined as an absolute neutrophil value < 1500 mm^3 within 30 days prior to screening.
* Acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV) positive, or previously diagnosed immunodeficiency with an absolute neutrophil count < 1000 cells/mm^3.
* Those who are positive for treponema pallidum antibodies and positive for rapid plasma reagin test (RPR).
* AAV9 neutralizing antibody titer > 1:50
* Subjects with a history of active tuberculosis or active or inactive TB infection at screening.
* 4 weeks prior to screening, or those who plan to receive a live (attenuated) vaccine during the trial.
* Those who smoked more than 20 cigarettes per day or habitually used nicotine-containing products in the 3 months prior to screening, drank more than 14 units of alcohol per week (1 unit of alcohol = 360mL of beer or 45mL of spirits or 150mL of wine with 40% alcohol content) or took alcohol-containing products 2 days before administration.
* The investigators believe that there are other conditions that would have an impact on intolerance to this treatment or endpoint evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) within 28 days of a single intracoronary infusion of JV001 | 28 days
  To evaluate the DLT occurred within 28 days after JV001 infusion
Incidence of adverse events and serious adverse events within 1 year of administration | 1 year
  To evaluate the safety of JV001 treatment

SECONDARY OUTCOMES:
Left ventricular ejection fraction | Baseline, Week 12, Week 26, Week 52
  Changes in left ventricular ejection fraction (LVEF as percentage) as assessed by echocardiography
Myocardial remodeling assessed by Cardiac Magnetic Resonance (CMR) Imaging | Baseline, Week 26
  Changes in left ventricular mass (absolute (ml) and index (ml/m2). Changes in left ventricular diastolic volume (ml). Changes in right ventricular diastolic volume (ml). Changes in left ventricular stroke volume
Change in N-terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) from baseline to Week 2, 4, 12, 26, 52 | Baseline, Week 2, Week 4, Week 12, Week 26, Week 52
  To evaluate the changes in NT-proBNP of subjects at 2, 4, 12, 26, and 52 weeks after medication from baseline. NT-proBNP is a biomarker for heart failure with a higher level indicating increased mortality and cardiovascular hospitalization in patients with heart failure.
Change in 6-minute Walk Test (6MWT) from baseline to Week 12，26，52 | Baseline, Week 12, Week 26, Week 52
  The 6MWT measures the distance walked in meters during a 6-minute test. Lower scores compared to baseline indicate worsening in function, and higher scores compared to baseline indicate improvement in function.
Change in total immunoglobulin and neutralizing antibodies from baseline to Week 2, Week 4, Week 12, Week 26, Week 52 | Baseline, Week 2, Week 4, Week 12, Week 26, Week 52
  Evaluate the changes in the formation of Anti-AAV9 antibodies.
Change in vector DNA levels in subjects' biological samples from baseline to Day 1, Day2, Day7, Week 2, Week 4, Week 12, Week 26, Week 52 | Baseline, Day 1, Day2, Day7, Week 2, Week 4, Week 12, Week 26, Week 52
  To evaluate the changes of AAV viral load in subjects' biological samples from baseline
Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) score from baseline to Week 12，26，52 | Baseline, Week 12, Week 26, Week 52
  The MLHFQ is a patient-report questionnaire used to assess the quality of life of heart failure patients. Higher scores indicate a lower quality of life.
Change of New York Heart Association (NYHA) functional classification from baseline to Week 12，26，52 | Baseline, Week 12, Week 26, Week 52
  The NYHA functional classification is the most commonly used classification system for patients with heart failure. Changes from baseline to a higher class indicate a worsening in symptoms.

OTHER OUTCOMES:
Change in standard uptake value (SUV) of 18F-fluorodeoxyglucose-positron emission tomography (PET) imaging from baseline to Week 26. | Baseline, Week 26
  To evaluate the changes myocardial viability of subjects at 26 weeks after medication from baseline
Late gadolinium enhancement (LGE) by Cardiac Magnetic Resonance (CMR) Imaging | Baseline, Week 26
  To evaluate the changes myocardial fibrosis of subjects at 26 weeks after medication from baseline
Biomarkers for Heart Failure and Prognosis | Baseline, Week 2, Week 4, Week 12, Week 26, Week 52
  Change in growth stimulation expressed gene 2 (ST2, ng/ml) Change in Heart-type fatty acid binding protein (H-FABP, ng/ml) Change in High-sensitivity cardiac troponin (hs-cTn, ng/ml)
Change in Human procollagen Ⅲ propeptide (PⅢP) for cardiac fibrosis in blood samples | Baseline, Week 4, Week 12, Week 26, Week 52
  Human procollagen Ⅲ propeptide (PⅢP) is an indication of myocardial fibrosis.
Change in interleukin 1-beta (IL-1β) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-1β (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 2 (IL-2) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-2 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 4 (IL-4) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-4 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 5 (IL-5) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-5 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 6 (IL-6) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-6 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 8 (IL-8) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-8 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 10 (IL-10) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-10 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 12p70 (IL-12p70) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-12p70 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interleukin 17 (IL-17) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IL-17 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interferon-alpha (IFN-α) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IFN-α (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in interferon-gamma (IFN-γ) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  IFN-γ (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in tumor necrosis factor-alpha (TNF-α) measured using blood samples (pg/ml) | Baseline, Week 4, Week 12, Week 26, Week 52
  TNF-α (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in immunoglobulin A (IgA) measured using blood samples (g/L) | Baseline, Week 4, Week 12, Week 26, Week 52
  IgA (in g/L), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in immunoglobulin M (IgM) measured using blood samples (g/L) | Baseline, Week 4, Week 12, Week 26, Week 52
  IgM (in g/L), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Change in immunoglobulin G (IgG) measured using blood samples (g/L) | Baseline, Week 4, Week 12, Week 26, Week 52
  IgG (in g/L), an inflammatory marker, will be measured in blood samples to assess changes from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Schultheiss HP, Fairweather D, Caforio ALP, Escher F, Hershberger RE, Lipshultz SE, Liu PP, Matsumori A, Mazzanti A, McMurray J, Priori SG. Dilated cardiomyopathy. Nat Rev Dis Primers. 2019 May 9;5(1):32. doi: 10.1038/s41572-019-0084-1. PMID 31073128
- [Background] Chang ACY, Chang ACH, Kirillova A, Sasagawa K, Su W, Weber G, Lin J, Termglinchan V, Karakikes I, Seeger T, Dainis AM, Hinson JT, Seidman J, Seidman CE, Day JW, Ashley E, Wu JC, Blau HM. Telomere shortening is a hallmark of genetic cardiomyopathies. Proc Natl Acad Sci U S A. 2018 Sep 11;115(37):9276-9281. doi: 10.1073/pnas.1714538115. Epub 2018 Aug 27. PMID 30150400
- [Background] Sahin E, Colla S, Liesa M, Moslehi J, Muller FL, Guo M, Cooper M, Kotton D, Fabian AJ, Walkey C, Maser RS, Tonon G, Foerster F, Xiong R, Wang YA, Shukla SA, Jaskelioff M, Martin ES, Heffernan TP, Protopopov A, Ivanova E, Mahoney JE, Kost-Alimova M, Perry SR, Bronson R, Liao R, Mulligan R, Shirihai OS, Chin L, DePinho RA. Telomere dysfunction induces metabolic and mitochondrial compromise. Nature. 2011 Feb 17;470(7334):359-65. doi: 10.1038/nature09787. Epub 2011 Feb 9. PMID 21307849
- [Background] Wang D, Tai PWL, Gao G. Adeno-associated virus vector as a platform for gene therapy delivery. Nat Rev Drug Discov. 2019 May;18(5):358-378. doi: 10.1038/s41573-019-0012-9. PMID 30710128